CLINICAL TRIAL: NCT07178769
Title: Multicenter Randomized Open-label Controlled Clinical Study to Evaluate the Efficacy and Safety of a Nutritional Supplement Based on Bergamot, Artichoke and Other Ingredients After Four Months of Treatment in Reducing Cholesterol Levels in Patients With Moderate or Mild Hypercholesterolemia
Brief Title: Study To Evaluate The Efficacy And Safety Of A Nutritional Supplement Based On Bergamot, Artichoke And Other Ingredients For Reducing Cholesterol Levels In Patients With Hypercholesterolemia (Metachol+)
Acronym: METACHOL+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Arkopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METACHOL+; METACHOL+ (Other: Effice spi S.L.)
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-06

CONDITIONS: Cholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Gr 1) (Experimental): Patients being treated with a nutritional supplement based on bergamot, artichoke and other ingredients with one capsule every night at dinner with a glass of water for four months.
  Interventions: Dietary Supplement: ARKOSTEROL
- Arm 2 (Gr 2) (Experimental): Patients treated with a nutritional supplement based on bergamot, artichoke and other ingredients with two capsules every night at dinner with a glass of water for four months.
  Interventions: Dietary Supplement: ARKOSTEROL
- Arm 3 (Control): Patients not taking METACHOL+ (No Intervention): All patients in the study will be recommended to lead an active life and a healthy diet, providing them with instructions to follow according to their usual clinical practice.

INTERVENTIONS:
Dietary Supplement: ARKOSTEROL — After 2 and 4 months from the start of treatment, a follow-up will be carried out in which anthropometric data will be measured (weight, BMI, waist circumference), vital signs (blood pressure and pulse) and a sample will be taken for analysis to measure the following parameters: CT, LDL, HDL, triglycerides, VLDL, Apo A, Apo B, liver function (GOT, GPT) and kidney function (creatinine) and Liposcale ® (in case of treatment group).
  Arms: Arm 1 (Gr 1); Arm 2 (Gr 2)

SUMMARY:
The goal of this clinical trial with food supplement is to evaluate the effectiveness of a nutritional supplement based on bergamot, artichoke and other ingredients through low-density lipoprotein (LDL) values after four months of treatment compared to maintaining healthy lifestyle habits.

The secondary objectives are

* Evaluate the improvement of the lipid profile compared to maintaining healthy lifestyle habits.
* Evaluate the difference in effect between 1 tablet and 2 tablets daily in improving the lipid profile.
* Evaluate changes in anthropometric data and vital signs.
* Evaluate adherence to treatment
* Evaluate the safety profile of the product
* Evaluate satisfaction with treatment

There are three treatment arms:

1. Arm 1 (Gr 1): Patients being treated with a nutritional supplement based on bergamot, artichoke and other ingredients with one capsule every night at dinner with a glass of water for four months.
2. Arm 2 (Gr 2): Patients treated with a nutritional supplement based on bergamot, artichoke and other ingredients with two capsules every night at dinner with a glass of water for four months.
3. Arm 3 (Control): Patients not taking METACHOL+. All patients in the study will be recommended to lead an active life and a healthy diet, providing them with instructions to follow according to their usual clinical practice.

It is expected to recruit 207 patients in total, 69 in each group/arm

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing and able to understand and sign the informed consent after the nature of the study has been fully explained to them and they have passed the inclusion/exclusion criteria.
2. Patients aged greater than or equal to 18 years
3. Patients with moderate or mild cardiovascular risk, who have LDL levels greater than 130 mg/dl.

Exclusion Criteria:

1. Use of any other drug or food supplement for the treatment of hypercholesterolemia during the 30 days prior to selection.
2. Allergy or hypersensitivity to any of the components of the study treatment.
3. Decompensated cardiovascular disease, decompensated diabetes mellitus, decompensated HTN.
4. Serious medical conditions such as: cancer, serious chronic illness considered incompatible with participation in the study or others that may interfere with the study.
5. HIV-AIDS, Pregnancy or breastfeeding, occlusion of the central retinal artery (of foreseeable vascular origin), history of cardiovascular disease and familial hypercholesterolemia.
6. Liver, kidney or muscle disorders.
7. Psychiatric disorders or inability to sign the consent.
8. Subjects with extreme eating habits and/or with a significant history of anorexia nervosa, bulimia and other eating disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Difference in the change in LDL cholesterol after four months of treatment compared to the baseline visit between patients treated | four months
  Difference in the change in LDL cholesterol after four months of treatment compared to the baseline visit between patients treated with a nutritional supplement (regardless of its dose) and patients in the control group.
  Difference in the change in LDL cholesterol after four months of treatment compared to the baseline visit between patients in group 1, group 2 and patients in the control group.
Difference in the change in LDL cholesterol after fou months of treatment compared to the baseline visit between patients treated in 1, 2 and control group | four months
  Difference in the change in LDL cholesterol after four months of treatment compared to the baseline visit between patients in group 1, group 2 and patients in the control group

SECONDARY OUTCOMES:
change in triglycerides | 2-4 months
  Difference in the change in triglycerides after 2 and 4 months of treatment compared to the baseline visit between patients in group 1 and patients in group 2.
change in VLDL | 2-4 months
  Difference in the change in VLDL after 2 and 4 months of treatment compared to the baseline visit between patients in group 1 and patients in group 2
change in Apo A | 2-4 months
  Difference in the change in Apo A after 2 and 4 months of treatment compared to the baseline visit between patients in group 1 and patients in group 2.
change in Apo B | 2-4 months
  Difference in the change in Apo B after 2 and 4 months of treatment compared to the baseline visit between patients in group 1 and patients in group 2
change in Liposcale | 2-4 months
  Difference in the change in Liposcale after 2 and 4 months of treatment compared to the baseline visit between patients in group 1 and patients in group 2

CONTACTS AND LOCATIONS:
Overall Officials: Guyoux Aurelie, Study Director — Arkopharma Laboratories
Locations (6):
- Spain (6):
  - Centro de Salud Goya, Madrid, Madrid
  - Centro de Salud Daroca, Madrid, Madrid
  - Centro de Salud Avenida de Aragón, Madrid, Madrid
  - Centro de Salud Casco Antiguo, Cartagena, Murcia
  - Centro de Salud Isaac Peral, Cartagena, Murcia
  - Centro de Salud de Mazarrón, Mazarrón, Murcia

IPD SHARING:
Plan to Share IPD: No